CLINICAL TRIAL: NCT03212794
Title: Initiating Substance Use Disorder Treatment for Hospitalized Opioid Use Disorder Patients.
Acronym: ISTOP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Joji Suzuki, MD, Director, Division of Addiction Psychiatry, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2017P001036; 1K23DA042326-01A1 (NIH)
Record Dates: First submitted 2017-07-06; First posted 2017-07-11 (Actual); Results first posted 2023-12-26 (Actual); Last update posted 2023-12-26 (Actual); Status verified 2023-12

CONDITIONS: Opioid-use Disorder
MeSH Terms: conditions — Opioid-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): Subjects randomized to the experimental arm will be assigned to a recovery coach.In addition to being linked to a community buprenorphine or methadone treatment program, the recovery coach will work to meet weekly with the subject following discharge from the hospital to provide support.
  Interventions: Behavioral: Recovery coach
- Control (No Intervention): Subjects randomized to the control arm will receive treatment as usual. This means subjects are linked to ongoing outpatient treatment with buprenorphine or methadone.

INTERVENTIONS:
Behavioral: Recovery coach — The recovery coach will support the subjects in the following areas: 1) monitor and manage symptoms, 2) patient education and self-management, and 3) enlisting community and social supports. Encouragement to continue treatment will be a primary focus of the recovery coach. In addition, the coach will conduct weekly sessions on various topics and offer personal insights and facilitate a discussion.
  Arms: Experimental

SUMMARY:
The purpose of this 24-week study is to evaluate the impact of recovery coach intervention on rates of treatment retention, illicit opioid use, and readmission among hospitalized patients newly initiated on buprenorphine or methadone compared to the control intervention.

DETAILED DESCRIPTION:
Patients with opioid use disorder (OUD) frequently utilize hospitals due to soft tissue infections and other conditions that require inpatient level of care. Prior studies have indicated that OUD patients are often amenable to initiating buprenorphine treatment and can be successfully linked to outpatient treatment. However, hospitalized OUD patients initiated on buprenorphine have much lower treatment retention rates at 6-months compared to OUD patients initiating treatment in the outpatient setting. As such, there is a great need to identify strategies to improve treatment retention in this patient population. There is a growing body of evidence for the benefits of recovery coaches, who provide peer-delivered support services in the community. Tracing their origin to mutual support groups to supplement traditional clinical services, recovery coaches are individuals with lived experience of recovery. Studies of recovery coaches have demonstrated greater treatment retention, reduced substance use, and reduced inpatient utilization. However, no prior studies have examined the impact of recovery coaches in improving medication-assisted treatment retention. As such, the aim of this 24-week study is to evaluate the impact of recovery coach intervention on rates of treatment retention, illicit opioid use, and readmission among hospitalized patients newly initiated on buprenorphine or methadone compared to the control intervention. Patients who are successfully initiated on buprenorphine or methadone, and are willing to engage in treatment after discharge, will be eligible to enroll. Assessments will be conducted at baseline, 4 weeks, 12 weeks, and 24 weeks.

ELIGIBILITY:
Inclusion Criteria:

* English speaking, adults aged 18-75
* Diagnostic and Statistical Manual of Mental Disorders, 5th edition (DSM-5) diagnosis of opioid use disorder, severe, actively using illicit opioids until the time of hospitalization
* Have a working telephone
* Can identify at least 2 individuals who can act as points of contact following discharge from the hospital
* Willing to engage in treatment (either a psychosocial treatment program AND/OR medication treatment with methadone or buprenorphine)

Exclusion Criteria:

* Liver function test >3x upper normal limit
* Pregnant
* Psychotic disorder, active suicidality or homicidality
* Condition likely to be terminal in 24 weeks such as cancer
* Unable to perform consent due to mental status
* Engaged in substance abuse treatment in the last month prior to admission

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2019-02-11 (Actual); Primary Completion 2021-12-30 (Actual); Study Completion 2021-12-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joji Suzuki, MD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Friedmann PD, Suzuki J. More beds are not the answer: transforming detoxification units into medication induction centers to address the opioid epidemic. Addict Sci Clin Pract. 2017 Nov 15;12(1):29. doi: 10.1186/s13722-017-0092-y. No abstract available. PMID 29141667

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment for the study was conducted between February 2019 and December 2021 at Brigham and Women's Hospital, an urban academic hospital in Boston, Massachusetts.
Groups:
- Experimental: Subjects randomized to the experimental arm will be assigned to a recovery coach. In addition to being linked to a community buprenorphine or methadone treatment program, the recovery coach will work to meet weekly with the subject following discharge from the hospital to provide support.
  Recovery coach: The recovery coach will support the subjects in the following areas: 1) monitor and manage symptoms, 2) patient education and self-management, and 3) enlisting community and social supports. Encouragement to continue treatment will be a primary focus of the recovery coach. In addition, the coach will conduct weekly sessions on various topics and offer personal insights and facilitate a discussion.
Period: Overall Study
Arm/Group | Experimental | Control
Started | 16 | 13
Completed | 5 | 5
Not Completed | 11 | 8
Not completed — Participation terminated due to prolonged inpatient stay (never able to receive intervention). | 1 | 0
Not completed — Lost to Follow-up | 5 | 6
Not completed — Incarcerated; unable to participate | 2 | 0
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Death | 0 | 1
Not completed — Found to be ineligible after allocation | 0 | 1
Not completed — Relocated out of area | 2 | 0

BASELINE CHARACTERISTICS:
Population: Participants not analyzed were either workbook manual pilot subjects (n=2), investigator-terminated (n=1), or found to be ineligible after enrollment (n=1).
Groups:
- Total: Total of all reporting groups
Arm/Group | Experimental | Control | Total
Number analyzed (Participants) | 13 | 12 | 25
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 13 | 12 | 25
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.7 (10.1) | 46.1 (13.7) | 42.8 (12.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 4 | 8
  Male | 9 | 8 | 17
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 0 | 4
  Not Hispanic or Latino | 9 | 12 | 21
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 2 | 3
  White | 8 | 10 | 18
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 3 | 0 | 3
Education (highest level completed) [Count of Participants; unit: Participants]
  Primary school | 2 | 4 | 6
  Secondary school | 11 | 8 | 19
Marital status [Count of Participants; unit: Participants]
  Divorced / single / widowed | 9 | 9 | 18
  Married / living as a couple | 4 | 3 | 7
Work [Count of Participants; unit: Participants]
  Employed | 4 | 5 | 9
  Unemployed | 9 | 7 | 16
Psychiatric history [Count of Participants; unit: Participants]
  Major Depressive Disorder (MDD): History of diagnosis | 12 | 7 | 19
  Major Depressive Disorder (MDD): No history of diagnosis | 1 | 5 | 6
  Bipolar disorder: History of diagnosis | 1 | 3 | 4
  Bipolar disorder: No history of diagnosis | 12 | 9 | 21
  Attention Deficit Hyperactivity Disorder (ADHD): History of diagnosis | 4 | 3 | 7
  Attention Deficit Hyperactivity Disorder (ADHD): No history of diagnosis | 9 | 9 | 18
  Anxiety disorder: History of diagnosis | 6 | 5 | 11
  Anxiety disorder: No history of diagnosis | 7 | 7 | 14
  Post-traumatic stress disorder (PTSD): History of diagnosis | 7 | 5 | 12
  Post-traumatic stress disorder (PTSD): No history of diagnosis | 6 | 7 | 13
Substance use disorder history [Count of Participants; unit: Participants]
  Opioid use disorder: History of diagnosis | 13 | 12 | 25
  Opioid use disorder: No history of diagnosis | 0 | 0 | 0
  Tobacco use disorder: History of diagnosis | 12 | 7 | 19
  Tobacco use disorder: No history of diagnosis | 1 | 5 | 6
  Cocaine use disorder: History of diagnosis | 9 | 8 | 17
  Cocaine use disorder: No history of diagnosis | 4 | 4 | 8
  Amphetamine use disorder: History of diagnosis | 5 | 1 | 6
  Amphetamine use disorder: No history of diagnosis | 8 | 11 | 19
  Cannabis use disorder: History of diagnosis | 4 | 4 | 8
  Cannabis use disorder: No history of diagnosis | 9 | 8 | 17
  Alcohol use disorder: History of diagnosis | 7 | 5 | 12
  Alcohol use disorder: No history of diagnosis | 6 | 7 | 13
  Sedative/hypnotic use disorder: History of diagnosis | 4 | 2 | 6
  Sedative/hypnotic use disorder: No history of diagnosis | 9 | 10 | 19
Medication for opioid use disorder (MOUD) initiated during hospitalization [Count of Participants; unit: Participants]
  Buprenorphine | 8 | 5 | 13
  Methadone | 5 | 7 | 12

OUTCOME MEASURES:

1. Primary Outcome: Treatment Retention
Description: Primary outcome was retention in MOUD treatment at 6-months after discharge. If referred to programs affiliated with Brigham and Women's Hospital (BWH), the electronic health records were used to confirm treatment retention. Otherwise, retention was determined through self-report or confirmation with collateral contacts. If the electronic health record was not available for confirmation and the participant was lost to follow-up, the missing data was imputed as discontinuation of MOUD treatment.
Time Frame: 24 weeks after baseline
Population: All enrolled participants were included in analyses, apart from the workbook manual pilot subjects (n=2), the investigator-terminated participant (n=1), and the participant found to be ineligible after enrollment (n=1).
Measure: Count of Participants; unit: Participants
Arm/Group | Experimental | Control
Number analyzed (Participants) | 13 | 12
Participants | 5 | 5
Statistical Analysis 1: Comparison: Experimental vs Control; Test type: Superiority; p = 0.87, Chi-squared — Threshold for significance p<0.05

2. Secondary Outcome: Readmissions
Description: Percentage of participants experiencing hospital readmission at 6 months. The electronic health records were used to establish hospital readmission.
Time Frame: 24 weeks after baseline
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Experimental | Control
Number analyzed (Participants) | 13 | 12
Participants | 6 | 5
Statistical Analysis 1: Comparison: Experimental vs Control; Test type: Superiority; p = 0.82, Chi-squared — Threshold for significance p<0.05

3. Secondary Outcome: Days to Treatment Discontinuation
Description: Number of days until MOUD treatment discontinuation. If referred to programs affiliated with BWH, the electronic health records were used to confirm treatment retention. Otherwise, retention was determined through self-report or confirmation with collateral contacts. If the electronic health record was not available for confirmation and the participant was lost to follow-up, the missing data was imputed as discontinuation of MOUD treatment.
Time Frame: 24 weeks after baseline
Population: Also excluded are the workbook manual pilot subjects (n=2), the investigator-terminated participant (n=1), and the participant found to be ineligible after enrollment (n=1). Only individuals who discontinued treatment during the study are included in this analysis. In the experimental group, 4 individuals did not discontinue treatment. In the control group, 5 individuals did not discontinue treatment. A total of 9 individuals are excluded, Of those analyzed: Experimental: 9; Control: 7
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Experimental | Control
Number analyzed (Participants) | 9 | 7
Days | 59.11 (64.25) | 26.71 (30.91)
Statistical Analysis 1: Comparison: Experimental vs Control; Test type: Other; p = 0.92, Log Rank — Threshold for significance p<0.05; If no event occurred, the data from those individuals were right censored

4. Secondary Outcome: Days to Hospital Readmission
Description: Number of days until hospital readmission. Electronic health records were used to establish hospital readmission.
Time Frame: 24 weeks after baseline
Population: Excluded participants are workbook manual pilot subjects (n=2), the investigator-terminated participant (n=1), and the participant found to be ineligible after enrollment (n=1). Only individuals who had a hospital readmission are included in this analysis. In the experimental condition, 6 individuals did not have a readmission. In the control condition, 6 individuals did not have a readmission, leaving a total of 13 people to be analyzed (Experimental: 7; Control :6).
Measure: Median (Standard Deviation); unit: Days
Arm/Group | Experimental | Control
Number analyzed (Participants) | 7 | 6
Days | 72.57 (43.14) | 67.67 (54.46)
Statistical Analysis 1: Comparison: Experimental vs Control; Test type: Other; p = 0.85, Log Rank — Threshold for significance p<0.05; If no event occurred, the data from those individuals were right censored

ADVERSE EVENTS:
Time Frame: 6 months following each participant's initial hospital discharge
Arm/Group | Experimental | Control
All-Cause Mortality (participants affected / at risk) | 0/13 | 1/12
Serious Adverse Events (participants affected / at risk) | 6/13 | 7/12
Other Adverse Events (participants affected / at risk) | 0/13 | 0/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Experimental (N=13) | Control (N=12)
Death (General disorders) | 0 (0) | 1 (1)
Hospitalization - acute kidney injury (Renal and urinary disorders) | 1 (1) | 1 (1)
Hospitalization - bacteremia (General disorders) | 1 (2) | 1 (1)
Hospitalization - opioid overdose (Psychiatric disorders) | 1 (1) | 0 (0)
Hospitalization - abdominal bleed (Vascular disorders) | 0 (0) | 1 (1)
Hospitalization - infected total knee replacement (Infections and infestations) | 0 (0) | 1 (2)
Hospitalization - surgical fixation status post osteoarthritis (Surgical and medical procedures) | 1 (1) | 0 (0)
Hospitalization - cellulitis (Skin and subcutaneous tissue disorders) | 2 (2) | 2 (2)
Hospitalization - splenic rupture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Hospitalization - endocarditis (Infections and infestations) | 0 (0) | 1 (2)
hospitalization - acute on chronic back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
hospitalization - abdominal pain (General disorders) | 0 (0) | 1 (1)
hospitalization - spinal epidural abscess (Infections and infestations) | 0 (0) | 1 (2)
hospitalization - substance-induced psychosis (Psychiatric disorders) | 1 (1) | 0 (0)
hospitalization - suicidal ideation (Psychiatric disorders) | 1 (3) | 0 (0)
hospitalization - septic arthritis (Infections and infestations) | 0 (0) | 1 (1)
hospitalization - acute on chronic congestive heart failure (Cardiac disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Pilot study with a small sample size. Because of the launch of a "bridge" clinic at the hospital briefly after trial initiation, participants in both treatment arms may have had access to peer support, potentially diluting the impact of the intervention. Self-report used to ascertain MOUD treatment retention when medical records were not available to be examined. Illicit opioid use after hospital discharge relied on self-report without any toxicologic confirmation.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-09-04): https://cdn.clinicaltrials.gov/large-docs/94/NCT03212794/Prot_SAP_000.pdf
  • Informed Consent Form (2021-07-13): https://cdn.clinicaltrials.gov/large-docs/94/NCT03212794/ICF_001.pdf